CLINICAL TRIAL: NCT07377110
Title: Understanding the Impact of Endoscopy Immersion Training in Regional Endoscopy Academies: is it Value for Money?
Brief Title: Endoscopy Immersion Study.
Status: Recruiting | Type: Observational
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24/108/GHT
Record Dates: First submitted 2025-09-30; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Training; Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- Endoscopy trainees who have received (or are soon to undertake immersion training

SUMMARY:
Endoscopy services are under significant pressure and endoscopy training academies and immersion training are under review at a national level. To date, there has been no comprehensive evaluation of the different approaches to immersion training or a large-scale study looking at its impact on trainees and/or endoscopy services. The purpose of this study is to perform a process, impact and economic evaluation of current immersion training practices to determine if they are impactful and value for money.

DETAILED DESCRIPTION:
Retrospective quantitative analysis involves endoscopists (training between January 2022 and the study start date) who may (or may not) have undertaken immersion training. Prospectively analysis will be performed to evaluate the impact of immersion training.

ELIGIBILITY:
Inclusion Criteria:

Endoscopy trainees (Surgical, Gastroenterology or CE) who have received (or are soon to undertake) immersion training in either gastroscopy or colonoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Endoscopy trainees
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Rate of improvement in DOPS (Direct Observation of Procedural Skills) score during immersion training compared to base hospital training | 6 months from start of data collection
  Rate of change in DOPS supervision assessment overall score - % of ratings competent for independent practice. Case matched interrupted time series analysis immersion trainees versus non-immersion trainees.
Caecal intubation rate (CIR)/ duodenal (D2) intubation rate improvement during immersion training compared to base hospital training? | 6 months from start of data collection
  % of procedures where trainee endoscopist advances the whole length of the colon to the caecum / successful intubation of the second part of the duodenum (D2) without assistance. Case matched interrupted time series analysis immersion trainees versus non-immersion trainees.
Improvement in time, and number of procedures, required for certification during immersion training compared to base hospital training? | 6 months from start of data collection
  Number of days between starting training and achieving certification (allowing for breaks in training e.g. parental leave) and number of procedures performed between starting training and achieving full certification. Case matched interrupted time series analysis immersion trainees versus non-immersion trainees.
Increase in number of endoscopies performed independently post certification following immersion training compared to base hospital training? | 6 months from start of data collection
  Number of endoscopies performed independently 3 months / 6 months/ 12 months post-certification. Case matched interrupted time series analysis immersion trainees versus non-immersion trainees.
Improvement in confidence scores following immersion training. | 6 months from start of data collection
  Do trainees feel more confident following immersion training? Survey and/or in-depth interviews with immersion trainees.

CONTACTS AND LOCATIONS:
Locations (1):
- Gloucestershire Royal Hospital, Gloucester, Gloucestershire, United Kingdom